CLINICAL TRIAL: NCT06591949
Title: Investigation of the Effectiveness of Cognitive Exercise Therapy Approach (BETY) in Juvenile Idiopathic Arthritis
Brief Title: Cognitive Exercise Therapy Approach (BETY) in JIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Orkun Tüfekçi, Principal Investigator, PT, PhD(c), Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBA 24/1113
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Childhood Rheumatic Diseases; Juvenile Idiopathic Arthritis (JIA); Exercise
Keywords: Childhood rheumatic diseases; biopsychosocial model; BETY; Cognitive exercise therapy approach; Exercise
MeSH Terms: conditions — Arthritis, Juvenile; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BETY session group (Active Comparator): JIA patients participating in BETY sessions.
  Interventions: Other: BETY
- Control Group (Active Comparator): JIA patients followed up with a home exercise program.
  Interventions: Other: Control group

INTERVENTIONS:
Other: BETY — The cognitive Exercise Therapy Approach (Bilişsel Egzersiz Terapi Yaklaşımı-BETY) will be applied for 24 one-hour sessions, two days a week.
  Arms: BETY session group
Other: Control group — Control group will be followed up with a home exercise program, and notes will be taken.
  Arms: Control Group

SUMMARY:
Cognitive Exercise Therapy Approach (*Bilişsel Egzersiz Terapi Yaklaşımı*-BETY), an innovative method developed for adults with rheumatism, aims to promote behavioral change and prevent social isolation by focusing on exercises that provide pain management and functional gains. BETY also recognizes the importance of family education in achieving these goals. However, there is a need for studies on exercise approaches that fit the biopsychosocial model, such as BETY in childhood rheumatic diseases.

BETY is an innovative exercise approach based on the biopsychosocial model that aims to change the patient's cognitions through exercise, specifically developed for patients with rheumatism. This approach includes function-oriented trunk stabilization exercises, chronic pain management, and authentic dance therapy training targeting positive cognitive displacement. It is carried out in a routinized structure that continues for years on a face-to-face basis in groups and individually.

Interventions that provide physical and psychosocial support are needed in childhood rheumatic diseases. Learning to exercise the muscles surrounding the joints at the proper traction angle through exercise with BETY, gaining the ability to manage chronic pain during the day, gaining positive cognitive displacement skills, and having the opportunity to socialize through both individual and group exercises constitute the basis of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with JIA,
* Aged between 7 and 18,
* Individuals who volunteered to participate in the study.

Exclusion Criteria:

* Patients with advanced heart/lung/liver/kidney disease, neurologic disease and malignancies,
* Individuals who have undergone major orthopedic surgery.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Juvenile Arthritis Biopsychosocial Questionnaire-JAB-Q-Patient | Three months
  Developed in 2018 in Turkey, it is a patient/parent-centered measurement method that helps to evaluate the biopsychosocial aspects of the patient, such as disease activity, posture, functional and psychosocial status, fatigue, performance at school. The results obtained from a total of 33 questions are used to evaluate the functional status of children, while their psychosocial status is recorded according to their answers to 21 questions. Scored between 0-164. A high score indicates a poor psychosocial status.
Juvenile Arthritis Biopsychosocial Questionnaire-JAB-Q-Family | Three months
  JAB-Q is used to assess the biopsychosocial status of patients and their parents. JAB-Q is a multidimensional questionnaire with a parent (family) form. The questionnaire developed in Turkish is completed by one of the parents/persons responsible for the child. The family form assesses the biopsychosocial status of the parent from their perspective and scores between 0 and 38. Higher scores indicate worse biopsychosocial status.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale - Parent Version (PCS-P) | Three months
  It is assessed with a 5-point Likert scale ranging from 0 (never) to 4 (always) and consists of 13 items. Parallel to the child questionnaire, it assesses three domains: rumination, magnification, and helplessness. A total score between 0-52 is obtained; higher scores reflect a higher level of catastrophizing in parents.
Child and Adolescent Scale of Participation (CASP): | Three months
  It is a 20-question questionnaire that evaluates the community participation of children and adolescents in school, neighborhood, and close environments. The questionnaire includes four sub-sections: 6 questions about home participation, four about neighborhood and community participation, five about school participation, and five about home and community participation. The questionnaire rating is expected by age (full participation), somewhat limited, very limited, not applicable, and not applicable. The family of the child or primary carer completes the questionnaire. The person completing the questionnaire is asked to select the answer that best describes the participation of a child in their care. As a result, the assessment is based between 0-100 points, with higher scores describing a better level of involvement.
Childhood Health Assessment Questionnaire (CHAQ) | Three months
  The CHAQ assesses the functional abilities of children with JIA in activities of daily living. It consists of eight subsections (dressing and personal care, standing up, eating, walking, body care, reaching, holding, and activities). It also assesses pain and general well-being with a visual analog scale. Scores range between 0 and 3 points. A high score is an indicator of low functionality.
Pain Catastrophising Scale-Child (PPS-C) | Three months
  It consists of 13 items describing different thoughts and feelings that children may experience when they feel pain. The questionnaire measures three areas: rumination, magnification, and helplessness. All items are evaluated on a 5-point Likert scale ranging from 0 (never) to 4 (always). Higher scores indicate more catastrophic pain beliefs. The total score is scored between 0 and 52.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Will not be shared to protect the data of individuals